CLINICAL TRIAL: NCT05679648
Title: Evaluation of Hepatic Steatosis and Fibrosis in Rheumatoid Arthritis Patients: a Cross-sectional Case-control Study
Brief Title: Hepatic Steatosis and Fibrosis in Rheumatoid Arthritis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amr Hamed, Lecturer, Sohag University
Other Study IDs: Soh-Med-22-11-17
Record Dates: First submitted 2022-12-25; First posted 2023-01-11 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Hepatic Steatosis and Fibrosis in Rheumatoid Arthritis Patients
Keywords: hepatic steatosis; rheumatoid arthritis
MeSH Terms: conditions — Fatty Liver; Arthritis, Rheumatoid | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid arthritis patients
  Interventions: Diagnostic Test: ultrasonography
- control
  Interventions: Diagnostic Test: ultrasonography

INTERVENTIONS:
Diagnostic Test: ultrasonography — studying degree of steatosis

SUMMARY:
studying the prevalence of hepatic steatosis and fibrosis in a large scale of patients with RA and healthy controls

ELIGIBILITY:
Inclusion Criteria:

1. RA according to the American College of Rheumatology (ACR)/EULAR 2010 criteria (Aletaha et al., 2010)
2. Age≥18 years

Exclusion Criteria:

* History of hepatitis B and C virus infection.
* Receiving hepatotoxic drugs other than RA-specific drugs.
* Alcohol abuse (i30 g/day in men and ⩾20 g/day in women).
* Diagnosis of Wilson's disease, α1-antitrypsin deficiency or hemochromatosis.
* Autoimmune liver disease.
* Cancer.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The outpatient clinic of the Rheumatology Department in Sohag University
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
degree of hepatic steatosis | 1 day during examination
  degree of hepatic steatosis by ultrasonography and Hepatic Steatosis Index.
degree of hepatic fibrosis | 1 day during examination
  degree of hepatic fibrosis by FIB-4 and APRI tests

IPD SHARING:
Plan to Share IPD: No